CLINICAL TRIAL: NCT06180304
Title: Examine the Effects of 24-week Exercise Program on Functional Capacity, Cognitive Capacity, and Quality of Life in Individuals With Intellectual and Developmental Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Politécnico de Leiria (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: FitnessParaAMente
Record Dates: First submitted 2023-11-27; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Intellectual Disabilities
MeSH Terms: conditions — Intellectual Disability | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Indoor training group (Experimental): Exercise group in a gym.
  Interventions: Other: Exercise training
- outdoor training group (Experimental): Exercise group in an outdoor space.
  Interventions: Other: Exercise training
- Control group (No Intervention): No exercise group.

INTERVENTIONS:
Other: Exercise training — The indoor physical exercise program was carried out in a gym with weight machines. The physical exercise program was divided into four parts. Part I: playful game or shuttle run (5 to 7 minutes). Part II: aerobic training (treadmill; 10 minutes; 40% to 80% of Heart Rate Reserve; between 12 to 17 according to the Borg Rating Of Perceived Exertion Scale; between 5 to 8 according to the Borg Category-Ratio 10 Scale. Part III: strength training (more or less 25 minutes; Leg Press + Chest Press + Leg Extension + Lat Pull Down + Leg Curl + Shoulder Press; 40-80% of 3 maximum repetitions; 10-15 reps; 2-3 sets). Part IV: 4 static stretches (30 to 60 seconds each).
  Arms: Indoor training group; outdoor training group

SUMMARY:
Physical inactivity and a sedentary lifestyle are prevalent in the population with intellectual and developmental disabilities, and they do not comply with the World Health Organisation's physical activity guidelines. Due to physical inactivity and a sedentary lifestyle, these individuals have low levels of physical fitness (decreasing functional capacity and success in carrying out activities of daily living), with an increased risk of acquiring other comorbidities such as type II diabetes, hypertension, cholesterol and metabolic syndrome, affecting their quality of life.

One of the reasons found in the literature for physical inactivity and sedentary lifestyles in individuals with intellectual and developmental disabilities is the existence of barriers that prevent/difficulty their practice, namely the lack of adapted physical exercise programmes, limited financial resources and lack of venues for their practice. Consequently, there is a dearth of research, including little clarity on the intervention protocols used and a variety of methodologies that address the applicability of non-pharmacological, psychological and psychosocial interventions, such as physical exercise programmes, for the promotion of various variables.

One of the most studied relationships is between exercise and the promotion of physical fitness, confirming its direct impact on functional capacity. Bearing in mind that studies on cognitive decline only assess some variables that may be associated but do not represent it on their own, such as attention, memory and language fluency. With regard to quality of life, an 8-week multidisciplinary exercise intervention programme aimed to improve quality of life, professional and peer support for activity, abdominal strength and metabolic equivalent gait of the tasks, however, the physical exercise programme is unclear and multimodal. On the other hand, a previous systematic review associated the effects of physical exercise with variables related to quality of life, namely pain, general health and anxiety. In studies focusing on physical activity, these variables have been shown to be predictors of quality of life, however, studies with physical exercise programmes are still cautious or unclear.

Thus, alternative and innovative solutions to promote/maintain physical function, reduce the risk of onset of cognitive decline in early life and promote/maintain the quality of life of individuals with Intellectual and Developmental Difficulty should include physical exercise. Taking this introductory approach into account, this non-randomised experimental study aimed to analyse the effects of two 24-week physical exercise programmes (indoor and outdoor) on functional capacity, cognitive decline and quality of life in institutionalised individuals with intellectual and developmental disabilities.

ELIGIBILITY:
Adult institutionalized volunteers from Leiria region (Center Portugal) participated in the exercise intervention program.

Participants were selected using the following inclusion criteria:

* adults with IDD;
* without medical contraindications;
* age over 18 years;
* with mild, moderate or severe IDD diagnosis (Down Syndrome inclusive);
* success in performing movements such as pulling/pushing;
* ability to carry out the intended assessments.

Additionally, we also used the following exclusion criteria:

* individuals who cannot commit for 6 months;
* individuals with other associated pathologies;
* contraindications to PE;
* inability to walk unassisted;
* profound IDD;
* inability to communicate;
* non-delivery of the duly signed informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Changes in Quality of Life | week 0 and 24
  The Portuguese version of the Personal Outcomes Scale was used. The instrument was applied by technicians with specific training aiming to evaluate QoL in people with IDD. The Personal Outcomes Scale includes eight domains, each containing five questions, making a total of forty questions, presented with three response options, through the Likert format, and a higher score (points) indicates better QoL (e.g., 3 = always; 2 = sometimes; 1 = seldom or never). For self-report measure, all composite reliability coefficients were within standards for acceptable internal consistency ranging from 0.75 to 0.91.
Changes in Cognitive function | week 0 and 24
  The Mini-Mental State Examination (MMSE) is a simple paper and pencil test with an easy and quick application (about 5 to 10 minutes) aiming to screen cognitive decline. MMSE test was adapted to the Portuguese population by Guerreiro et al. (1994) and used with IDD population. The thirty items questionnaire (scored 0 value - when the person gives an incorrect answer or simply does not answer or scored 1value - when the person answers correctly), is organized in six domains: Orientation, Retention, Attention and Calculation, Evocation, Language. The maximum test score is thirty points, with higher scores indicating better results. Its score ranges from 0 to 30 points, and the cut-off values that classify individuals into cognitive profiles are: a) severe cognitive impairment (1-9 pts); b) moderate cognitive impairment (10-18 pts) mild cognitive impairment (19-24 pts), d) normal cognitive status (25 pts and above).
Changes in Functional Capacity | week 0, 12 and 24
  Fullerton battery of functional tests was used to assess physical fitness, namely:
  i) the "sit to stand" for 30 seconds test, validated for the IDD population evaluated the strength and resistance of the lower limbs. The purpose of the test is to assess the strength and the resistance of the lower limbs (number of executions in 30 seconds without using the upper limbs - repetitions). The test begins with the participant sitting in the middle of the chair, with the back straight and feet shoulder-width apart and fully supported on the floor;
  ii) the "Timed up and Go" test, validated for the IDD population aimed to assess physical mobility, namely speed, agility and dynamic balance (seconds);
  iii) the "6-minute walk" test validated for IDD population aimed to assess aerobic resistance by covering the greatest distance in 6 minutes (minutes).

CONTACTS AND LOCATIONS:
Locations (1):
- Miguel Jacinto, Coimbra, Portugal